CLINICAL TRIAL: NCT06430086
Title: Mechanistic Effect of Walnut Consumption on Sleep Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); California Walnut Commission (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAV1362; GRANT13949102 (Other Grant/Funding Number: USDA/NIFA)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Poor Sleep Quality
Keywords: Randomized crossover study; Controlled feeding; Dietary intervention; Inpatient visit; Outpatient monitoring

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Who Masked: Investigator
Masking Description: Statistician will be masked to study condition. Participants cannot be masked. Other personnel involved in the study cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut - washout - HCHS (Experimental): Participants will consume 3 servings/day of walnuts (3 oz/d) over 4 days and have a washout for 2-3 weeks then crossover to consume 3 equicaloric servings of a HCHS food over 4 days.
  Over each 4-day period, participants will sleep and eat at home for the first 3 days and will be admitted to the Inpatient Clinical Research Resource of the Irving Institute for Clinical and Translational Research of CUIMC on day 4 for in-depth profiling circadian physiology. Participants will be discharged on the morning of day 5.
  Interventions: Other: Walnut consumption; Other: HCHS consumption
- HCHS - washout - Walnut (Experimental): Participants will consume 3 equicaloric servings of a HCHS food over 4 days and have a washout for 2-3 weeks then crossover to consume 3 servings/day of walnuts (3 oz/d) for 4 days.
  Over each 4-day period, participants will sleep and eat at home for the first 3 days and will be admitted to the Inpatient Clinical Research Resource of the Irving Institute for Clinical and Translational Research of CUIMC on day 4 for in-depth profiling circadian physiology. Participants will be discharged on the morning of day 5.
  Interventions: Other: Walnut consumption; Other: HCHS consumption

INTERVENTIONS:
Other: Walnut consumption — Participants will add one serving (1 oz) of walnuts at their self-defined breakfast, lunch, and dinner for 4 days. The study will provide study foods at 3 main meals each day to evaluate a temporal effect of the food on melatonin concentrations throughout the day.
Other: HCHS consumption — Participants will add one HCHS food (one PopTarts® pastry) to each of their 3 main meals of the day for 4 days. The study will provide study foods at 3 main meals each day to evaluate a temporal effect of the food on melatonin concentrations throughout the day.
  An energy-matched high-carbohydrate, high-sugar (HCHS) alternative, representative of a common US snack food, on sleep quality in adults with habitually poor sleep quality.

SUMMARY:
Poor sleep quality is very common in modern society. Walnuts contain many nutrients that may be helpful for sleep, including melatonin and polyphenols. Some studies show that eating foods high in melatonin and polyphenols improves sleep quality, but walnuts have not been studied specifically. This study proposes to test if eating walnuts improves sleep compared to a food that lacks these sleep-promoting factors. The investigators expect that walnut consumption for 4 days will increase melatonin levels and lead to better sleep quality compared to a high-carbohydrate, high-sugar food. The study will enroll middle-aged and older adults with sleep complaints to participate in this study. Each person will eat the two different foods for 4 days each in random order. The 4-day periods will be separated by at least 2-3 weeks. Sleep quality will be measured by questionnaire and with a wrist monitor every day. The investigators will also do a sleep study using electroencephalography (EEG) on night 3 and take measures of circadian physiology (natural body rhythms) in the laboratory on day 4 (including overnight) by measuring body temperature and blood and urine melatonin. The study findings may provide new options to improve sleep health from increased walnut consumption.

DETAILED DESCRIPTION:
Walnuts are a nutrient-rich food which provides melatonin and polyphenols. While there is evidence that dietary intakes of foods high in melatonin and polyphenols positively influence sleep quality, the effect of walnuts has not been investigated. The investigators propose to fill this knowledge gap by testing the effects of walnut consumption on serum melatonin and resulting sleep and circadian biology. The study hypotheses are that walnut consumption for 4 days will increase melatonin levels, suggestive of more robust circadian rhythms, and lead to better sleep quality compared to a high-carbohydrate high-sugar (HCHS) equivalent. Using a randomized controlled crossover trial, the study aims to: 1) determine the effect of walnut vs HCHS consumption on melatonin levels; and 2) determine the effect of walnut vs HCHS consumption on sleep and circadian physiology. Adult males and females with poor sleep quality will consume three servings/day of walnuts or an equicaloric HCHS food for 4 days. Sleep quality will be measured nightly using the Karolinska Sleep Diary and wrist actigraphy; sleep architecture from polysomnography will be measured on night 3. Circadian physiology will be assessed on day 4 using body temperature and hourly serum melatonin and on the morning of day 5 from overnight urinary 6-sulfatoxymelatonin. Given the extent of poor sleep, our findings may open new avenues to improve sleep health from increased walnut consumption.

ELIGIBILITY:
Inclusion Criteria:

* Equal numbers of men and women (12 male and 12 post-menopausal female)
* Equal number of individuals with normal weight (18.5-24.9 kg/m2) and overweight (25-29.9 kg/m2)
* Participants will self-report poor sleep quality, reflected by a global score >5 on Pittsburgh Sleep Quality Index

Exclusion Criteria:

* Diagnosed sleep disorder
* Participants with conditions that could affect sleep will be excluded:

  * smoking, excessive caffeine intake (>300 mg/day)
  * shift work
  * chronic pain
  * diagnosis of a chronic disease (e.g., uncontrolled hypertension, pre-diabetes, type 2 diabetes, chronic kidney disease, chronic obstructive pulmonary disease),
  * autoimmune diseases
  * cardiovascular event or cancer in the past 24 months
  * psychiatric/neurologic disease or disorder, or sleep disorder (diagnosed or high risk for sleep apnea, chronic insomnia, restless leg syndrome, narcolepsy)
  * use of medications that influence CYP1A2 enzymes
* Allergy/intolerance to nuts, tree nuts, or unwilling to eat study foods

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum melatonin | Baseline (9AM; Hour 0), Hour 1, Hour 2, Hour 3, Hour 4, Hour 5, Hour 6, Hour 7, Hour 8, Hour 9, Hour 10, Hour 11, Hour 12, Hour 13, Hour 14, Hour 15 (Midnight)
  Serum melatonin will be measured via last testing of blood samples collected on day 4, in an inpatient setting. Repeated for each phase.
Sleep quality index | Night 1, Night 2, Night 3, Night 4
  Sleep quality will be assessed daily using wrist actigraphy. Variables include sleep fragmentation index and sleep efficiency. Repeated for each phase.
Slow wave sleep index | Night 3
  Slow wave sleep will be measured using electroencephalography, in the participant's home. Repeated for each phase.

SECONDARY OUTCOMES:
6-sulfatoxymelatonin level | Night 4 to morning of Day 5 (Approximately up to 12 hours)
  This is to measure Melatonin production in urine samples. Repeated for each phase.
Body temperature | Day 4
  Proximal to distal body temperature gradient measured using thermochron devices (iButtons). Repeated for each phase. In patient. Over 24 hours.
Sleep quality score | Days 2, 3, 4, 5
  Self-reported sleep quality assessed using the Karolinska Sleep Diary (higher score represents better sleep). Repeated for each phase.

OTHER OUTCOMES:
NFkB level | Day 4 (or Day 5)
  This is to measure Endothelial cell inflammation in endothelial cells collected from a forearm vein. Repeated for each phase. Fasted sample.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Associate Professor of Nutritional Medicine
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to Zenodo, a generalist repository that is participating in the NIH Generalist Repository Ecosystem Initiative. We will submit metadata associated with the datasets to Zenodo. The repository will provide metadata, persistent identifiers, and long-term access for open and controlled access. Each study created in Zenodo is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication. To request access of the data, researchers will use the standard processes at Zenodo. Given that we seek the widest possible availability, in most cases all that is necessary is obtaining a Zenodo account from the repository web site.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of final study completion.
URL: https://about.zenodo.org/policies/